CLINICAL TRIAL: NCT03804749
Title: A Randomized, Double-blind, Placebo-controlled, Single-dose, Dose-escalation Study to Evaluate the Tolerance and Pharmacokinetics of Suramin Sodium in Healthy Chinese Adults
Brief Title: Study to Evaluate the Tolerance and Pharmacokinetics of Suramin Sodium
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Guangdong Kangda Pharmaceutical Co., Ltd (Industry)
Responsible Party: Principal Investigator, shentu jianzhong, Ph.D.（Pharm）, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LC00-043
Record Dates: First submitted 2018-12-28; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Hand, Foot and Mouth Disease
Keywords: suramin sodium
MeSH Terms: conditions — Hand, Foot and Mouth Disease | interventions — Suramin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind, placebo control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1-1 (Experimental): The dose of suramin sodium is 10 mg/kg
  Interventions: Drug: suramin sodium
- Group 1-2 (Placebo Comparator): The placebo is 0.9% sodium chloride injection
  Interventions: Other: placebo
- Group 2-1 (Experimental): The dose of suramin sodium is 15mg/kg
  Interventions: Drug: suramin sodium
- Group 2-2 (Placebo Comparator): The placebo is 0.9% sodium chloride injection
  Interventions: Other: placebo
- Group 3-1 (Experimental): The dose of suramin sodium is 20mg/kg
  Interventions: Drug: suramin sodium
- Group 3-2 (Placebo Comparator): The placebo is 0.9% sodium chloride injection
  Interventions: Other: placebo

INTERVENTIONS:
Drug: suramin sodium — The trial will start from the low dose (10mg/kg) group, followed by the middle dose (15mg/kg) and high dose (20mg/kg) groups, only after the safety in the previous dose group has been demonstrated.。
  Arms: Group 1-1; Group 2-1; Group 3-1
Other: placebo — Placebo is 0.9% sodium chloride injection.
  Other Names: 0.9% sodium chloride injection
  Arms: Group 1-2; Group 2-2; Group 3-2

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single-dose with three incremental doses, Phase 1 study to evaluate the tolerance and pharmacokinetics of suramin sodium for injection in Chinese healthy adults.

DETAILED DESCRIPTION:
A total of 36 subjects are divided into three dosage groups: 10mg/kg, 15mg/kg and 20mg/kg, in which 20mg/kg is the conventional dosage per international pharmacopoeias for established indications of suramin sodium. Each dose group contains 12 subjects. By randomization, 10 of them receive suramin sodium while 2 of them receive placebo (0.9% sodium chloride injection）. The trial will start from the low dose (10mg/kg) group, followed by the middle dose (15mg/kg) and high dose (20mg/kg) groups, only after the safety in the previous dose group has been demonstrated.

All subjects in each dose group will be un-blinded after blood/urine collection and safety evaluation on Day 28. After that, blood and urine samples on suramin-dosing subjects will continue to collect on Days 56、84、112 and 140.

Subjects receiving placebo will complete the study on Day 28 if no AE is observed, or follow up till the adverse event (AE) return to normal or stabilize if AE is detected.

Blood and urine samples will be tested by a validated LC/MS method for pharmacokinetic study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers who fully understand the purpose, content, benefits and possible adverse reactions of the test and voluntarily sign written informed consent prior to the commencement of any test-related activities.
2. Healthy males or females, aged 18 to 45 years (including 18 and 45 years).
3. Male subjects weighed 50-75 kg (including 50 and 75 kg), female subjects weighed 45-75 kg (including 45 and 75 kg), body mass index (BMI) was 18.0-26.0 kg/m2 (including 18.0 and 26.0 kg/m2), where BMI = body weight (kg)/height2 (m2).
4. Have the ability to communicate with investigator and abide by the management regulations of the hospital and the clinical research.

Exclusion Criteria:

1. Fail in physical examination, vital signs measurement, standard 12-lead electrocardiogram, chest X-ray, laboratory examination [blood routine, urine routine, blood biochemistry, blood coagulation function, infectious diseases, blood pregnancy (only for women of childbearing age), as judged by the investigator to be of clinical significance.
2. With gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, immunity, mental or cardiovascular diseases.
3. Has allergic constitution (allergic to two or more substances), or allergic history, or known allergic to suramin sodium.
4. Cannot tolerate venipuncture and/or have a history of fainting blood or needle.
5. Has massive blood loss (> 400 mL) or had donated blood/blood components within the first six months of screening, or who planned to donate blood/blood components during the study period.
6. Had participated in clinical trials of drugs and took research drugs within three months before screening.
7. Smoke more than five cigarettes a day (including nicotine substitutes) or the same amount of tobacco products in the first three months of screening.
8. Has history of drug abuse within 5 years before screening, or those who had used drugs within 3 months before screening.
9. Has a history of alcoholism or moderate alcoholism in the first two years of screening (moderate alcoholism is defined as drinking more than 3 units per day or 21 units per week; a bottle of 350 mL beer, 120 mL white wine, 150 mL wine or 30 mL spirits is one unit).
10. Pregnant or lactating women, or subjects (or their partners) who have pregnancy plans during the trial and within three months after the end of the study, or who do not agree to use non-drug contraceptive measures during the trial.
11. Positive urine drug screening in screening stage.
12. Alcohol urine positive in screening stage.
13. Nicotine positive in screening stage.
14. With acute diseases in screening period.
15. Had used any prescription, over-the-counter, vitamin products or Chinese herbal medicines within 14 days before enrollment.
16. Female subjects of childbearing age who did not take non-drug contraceptive measures within 14 days before admission.
17. Not suitable for participating into the trial as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-12-19 (Actual); Primary Completion 2019-12-19 (Estimated); Study Completion 2020-12-19 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with adverse events | [ Day 1 to Day 140 ]
  Adverse events
the area under the plasma concentration-time curve (AUC) from time zero to the time of the last measurable concentration (AUC0-t) of suramin sodium | [ Day 1 to Day 140 after study drug administration ]
  Pharmacokinetics parameters
the AUC from time zero to infinity (AUC0-inf) of suramin sodium | [ Day 1 to Day 140 after study drug administration ]
  Pharmacokinetics parameters
maximum plasma concentration (Cmax ) of suramin sodium | [ Day 1 to Day 140 after study drug administration ]
  Pharmacokinetics parameters
half life （t1/2） of suramin sodium | [Day 1 to Day 140 after study drug administration ]
  Pharmacokinetics parameters
clearance （CL） of suramin sodium | [ Day 1 to Day 140 after study drug administration ]
  Pharmacokinetics parameters
apparent volume of distribution（Vd） of suramin sodium | [ Day 1 to Day 140 after study drug administration ]
  Pharmacokinetics parameters
the amount of drug excreted into the urine from time zero to time 7 days（Ae0-t） of suramin sodium | [ Day 1 to Day 7 after study drug administration ]
  Pharmacokinetics parameters

CONTACTS AND LOCATIONS:
Overall Officials: First Affiliated Hospital Zhejiang University, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No